CLINICAL TRIAL: NCT06893549
Title: Effect of Lactobacillus Plantarum GKK1 Supplementation on Anti-fatigue Health Effects
Acronym: GKK1-Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Principal Investigator, Chi-Chang Huang, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-24-034-A2; IRB-24-034-A2 (Other: Landseed Hospital International Institutional Review Board)
Record Dates: First submitted 2025-03-17; First posted 2025-03-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Exercise-Induced Fatigue; Muscle Fatigue; Sports Performance; Fatigue Recovery
Keywords: Probiotic Supplement; Exercise Fatigue; Lactiplantibacillus paraplantarum GKK1; Physical Performance; Muscle Damage; Recovery; Anaerobic Power; Explosive Power; Isometric Strength; Sports Nutrition

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, placebo-controlled parallel-group trial comparing the effects of Lactobacillus plantarum GKK1 supplementation with a placebo in healthy adults.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blind, meaning that the participants, care providers, investigators, and outcomes assessors are unaware of the assigned interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactobacillus plantarum GKK1 Probiotic Group (Experimental): Participants in this group will receive a daily oral supplementation of Lactobacillus plantarum GKK1 probiotic capsules for 28 days. Each capsule contains 50 billion CFU, with a total daily intake of 100 billion CFU. On Day 29, participants will undergo an exhaustive exercise test, and various physiological and biochemical markers will be assessed pre- and post-exercise.
  Interventions: Dietary Supplement: Lactobacillus plantarum GKK1 Probiotic
- Placebo Group (Placebo Comparator): Participants in this group will receive a daily oral supplementation of placebo capsules for 28 days. The placebo capsules contain microcrystalline α-cellulose, magnesium stearate, and silicon dioxide, with identical appearance and taste to the probiotic capsules. On Day 29, participants will undergo an exhaustive exercise test, and various physiological and biochemical markers will be assessed pre- and post-exercise.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum GKK1 Probiotic — Participants in the probiotic group will receive a daily oral supplementation of Lactobacillus plantarum GKK1 probiotic capsules for 28 days. Each capsule contains 50 billion CFU, with a total daily intake of 100 billion CFU. The probiotic strain Lactobacillus plantarum GKK1 has been selected for its potential benefits in reducing exercise-induced fatigue and enhancing physical performance. The supplementation period will be followed by an exhaustive exercise test to assess physiological and biochemical changes.
  Other Names: Probiotic Supplement
  Arms: Lactobacillus plantarum GKK1 Probiotic Group
Dietary Supplement: Placebo — Participants in the placebo group will receive a daily oral supplementation of placebo capsules for 28 days. The placebo capsules are identical in appearance, taste, and weight to the probiotic capsules but contain only microcrystalline α-cellulose, magnesium stearate, and silicon dioxide. The supplementation period will be followed by an exhaustive exercise test to assess physiological and biochemical changes.
  Other Names: Placebo Supplement
  Arms: Placebo Group

SUMMARY:
Title: Effect of Lactobacillus plantarum GKK1 Supplementation on Anti-Fatigue Health Effects: A Randomized, Double-Blind, Placebo-Controlled Trial

This study aims to investigate the effects of Lactobacillus plantarum GKK1 supplementation on fatigue reduction and physical performance enhancement in healthy adults. Probiotics are known to modulate gut microbiota and may influence exercise-induced fatigue and recovery.

A total of 48 healthy adults aged 18-35 years will be randomly assigned to either the probiotic group (Lactobacillus plantarum GKK1, 100 billion CFU/day) or the placebo group, with supplementation for 28 consecutive days. On Day 29, participants will perform an exhaustive exercise test, and their anaerobic power, explosive power, isometric muscle strength, and stress hormone levels (cortisol, catecholamines, GH, testosterone, hs-CRP) will be evaluated before and after exercise.

The primary objective is to assess whether probiotic supplementation can reduce exercise-induced fatigue and muscle damage while improving recovery performance. Blood biochemical markers, muscle damage indicators, and subjective fatigue perception will also be analyzed.

This study is conducted at National Taiwan Sport University, under ethical approval from Landseed Hospital IRB (IRB-24-034-A2).

DETAILED DESCRIPTION:
Probiotic supplementation has garnered increasing interest in sports science due to its potential effects on gut microbiota modulation, systemic inflammation, and exercise recovery. Lactobacillus plantarum GKK1, a strain isolated from fermented plant sources, exhibits promising antioxidative and anti-inflammatory properties, making it a candidate for supporting physical resilience and fatigue recovery in active individuals.

This study is designed as a randomized, double-blind, placebo-controlled clinical trial aiming to evaluate whether supplementation with L. plantarum GKK1 can attenuate physiological stress responses and muscle damage following exhaustive exercise in healthy adults. The probiotic intervention lasts for 28 consecutive days, during which participants maintain habitual dietary and lifestyle behaviors, except for the avoidance of other functional supplements.

The experimental exercise model includes a structured fatigue-inducing protocol involving repetitive plyometric movements. This model was selected to simulate high-intensity sport-like conditions while reliably inducing measurable muscle stress. Following this challenge, blood and urine samples are collected at predefined time points to monitor temporal changes in selected biochemical markers.

The trial incorporates both objective and subjective metrics, including validated physical performance tests and standardized fatigue perception scales. Biochemical assessments are conducted using automated clinical analyzers and immunoassay techniques under Good Laboratory Practice conditions. The core hypothesis posits that probiotic intervention will result in lower elevations in stress hormones and muscle damage biomarkers, along with improved physical performance maintenance compared to placebo.

All procedures are conducted at the National Taiwan Sport University under IRB approval (IRB-24-034-A2). This trial may provide evidence for the application of probiotic supplementation as a supportive strategy for fatigue management and exercise recovery enhancement in recreationally active populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 35 years
* Non-smokers and non-alcohol drinkers
* No history of chronic disease (e.g., cardiovascular disease, diabetes, asthma, metabolic disorders)
* No musculoskeletal injuries in the past 6 months
* Not taking anti-inflammatory or pain-relief medication in the past month
* No history of gastrointestinal surgery (excluding hernia or polyp removal)
* No allergies to dairy or probiotics

Exclusion Criteria:

* Diagnosed with cardiovascular, metabolic, or neurological disorders
* Regular consumption of probiotics within the last three months
* Pregnant or lactating women
* Individuals taking medication affecting hormonal balance or immune response
* Use of corticosteroids, NSAIDs, or muscle relaxants in the past month
* Participating in another clinical trial within the last three months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Change in Anaerobic Power | Time Frame: Day 0 (baseline), Day 29 before exercise, Day 29 three hours after exercise, and Day 30 twenty-four hours after exercise
  Anaerobic power will be assessed using a Wingate anaerobic test. Measurements include peak power (W/kg), average power (W/kg), and fatigue index (%). Higher values indicate better performance and lower fatigue.

SECONDARY OUTCOMES:
Change in Cortisol Levels | Day 0 (baseline), Day 29 before exercise, Day 29 three hours after exercise, and Day 30 twenty-four hours after exercise
  Serum cortisol levels (nmol/L) will be measured using enzyme-linked immunosorbent assay (ELISA). Cortisol is a biomarker of physiological stress and fatigue. Changes in cortisol concentration will be used to assess the participant's stress response to exhaustive exercise.
Change in Catecholamines Levels | Day 0 (baseline), Day 29 before exercise, Day 29 three hours after exercise, and Day 30 twenty-four hours after exercise
  Serum catecholamines (epinephrine, norepinephrine, and dopamine) will be measured using high-performance liquid chromatography (HPLC). These biomarkers reflect sympathetic nervous system activity and are associated with exercise-induced stress and fatigue.
Change in hs-CRP Levels | Day 0 (baseline), Day 29 before exercise, Day 29 three hours after exercise, and Day 30 twenty-four hours after exercise
  High-sensitivity C-reactive protein (hs-CRP) will be measured in serum (mg/L) using ELISA. hs-CRP is a marker of systemic inflammation and may increase in response to intense physical stress. This measurement helps assess the anti-inflammatory effect of probiotic supplementation.
Change in Creatine Kinase (CK) | Day 0 (baseline), Day 29 before exercise, Day 29 three hours after exercise, and Day 30 twenty-four hours after exercise
  Serum creatine kinase (CK) activity (U/L) will be assessed using an automated biochemical analyzer. CK is a widely used marker of muscle damage following intense exercise. Elevated levels may indicate muscle cell injury.
Change in Myoglobin Levels | Day 0 (baseline), Day 29 before exercise, Day 29 three hours after exercise, and Day 30 twenty-four hours after exercise
  Serum myoglobin (ng/mL) will be measured using a commercial assay kit. Myoglobin is released into the blood following muscle damage and is used as an early indicator of exercise-induced muscle injury.
Change in 3-Methylhistidine Levels | Day 0 (baseline), Day 29 before exercise, Day 29 three hours after exercise, and Day 30 twenty-four hours after exercise
  Urinary 3-methylhistidine concentration will be measured as a biomarker of muscle protein breakdown. The ratio of 3-methylhistidine to creatinine (μmol/mmol) will be used to assess muscle catabolism post-exercise.
Change in Subjective Fatigue Perception Score | Day 0 (baseline), Day 29 before exercise, Day 29 three hours after exercise, and Day 30 twenty-four hours after exercise
  Subjective fatigue perception will be assessed using a 10-point visual analog scale, where 0 indicates no fatigue and 10 indicates extreme fatigue. Participants will rate their perceived fatigue at specified time points to evaluate recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Sport University, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MC, Hsu YJ, Ho CS, Chang CH, Liu CW, Huang CC, Chiang WD. Evaluation of the Efficacy of Supplementation with Planox(R) Lemon Verbena Extract in Improving Oxidative Stress and Muscle Damage: A Randomized Double-Blind Controlled Trial. Int J Med Sci. 2021 May 3;18(12):2641-2652. doi: 10.7150/ijms.60726. eCollection 2021. PMID 34104096